CLINICAL TRIAL: NCT04573712
Title: FAME 1: The Effects of Apathy on Different Forms of Fatigue
Brief Title: The Effects of Apathy on Different Forms of Fatigue
Acronym: FAME1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-PP-20
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Apathy; Fatigue
MeSH Terms: conditions — Lethargy; Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue Severity Scale scores assessment (Experimental): Fatigue Severity Scale scores assessment
  Interventions: Other: Follow up and Assessment

INTERVENTIONS:
Other: Follow up and Assessment — each patient should wear an actigraph during a week and will be do some tests during 2hours (6min walk, apathy inventory, fatigue severity scale etc...)

SUMMARY:
60 participants with light neuro-cognitive disorders (30 apathetic, 30 non-apathetic) will be recruited from the CMRR (Centre Mémoire Ressources et Recherche) in Nice University Hospital and from the " Fragilily " Platform of the Nice University Hospital.

After verification by the investigator, if they meet the inclusion criteria and sign the informed consent, participants will have to wear an actigraph for one week in order to measure their level of activity.

Afterwards, participants will have to complete assessments and questionnaires to evaluate apathy (Apathy Motivation Index, Apathy Inventory), perceived fatigue (Fatigue Severity Scale, Borg scale), fatigability (6-min walking test, isometric strength test, double task), the stress level (Perceived Stress Scale) and depression (Geriatric Depression Scale).

Regarding the activity level, they will also be asked to perform tasks to evaluate their kinematic movements( through an actigraph), and their particular sensitivity towards effort and reward (through serious game 'Tap-piscine').

The total duration of the evaluation is a maximum of 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 65 and 85 years old coming for consultation at the RMC and the Fragility Platform
* DSM-5 diagnosis: minor neurocognitive disorders
* Subject must read and write in French.
* Subject must be registered in the national social security scheme.
* Ability to sign free and informed consent.

For the 'apathetic' group:

- Presence of apathy/emotional symptoms: at least 2 criteria according to the diagnostic criteria for apathy and a score higher than 8.5 in the MBI affective dimension.

For the 'non-apathetic' group:

- Absence of apathy/emotional symptoms: no criteria according to the diagnostic criteria for apathy and a score of less than 8.5 in the MBI affective dimension.

Exclusion Criteria:

* Motor or sensory disabilities likely to interfere with the tests.
* Presence of major psychiatric disorders (e.g., schizophrenia, major depressive episode, bipolar disorder)
* Patient under guardianship, curatorship or under legal protection

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
comparison of Fatigue Severity Scale scores between apathetic and non-apathetic subjects. | at inclusion
  the minimum score is 9 (worse outcome) and the maximum score is 63 (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PU-PH, Principal Investigator — CHU de NICE, Centre Mémoire Ressources et Recherches
Locations (1):
- Centre Memoire Ressources et Recherche, CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daumas L, Zory R, Robert P, Manera V. Apathetic patients with neurocognitive disorders are more fatigued and fatigable. Aging Clin Exp Res. 2022 Sep;34(9):2237-2241. doi: 10.1007/s40520-022-02146-4. Epub 2022 May 24. PMID 35608793